CLINICAL TRIAL: NCT01692119
Title: Pharmacy-based Interdisciplinary Program for Patients With Chronic Heart Failure (PHARM-CHF): A Randomized Controlled Trial
Brief Title: Pharmacy-based Interdisciplinary Program for Patients With Chronic Heart Failure
Acronym: PHARM-CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Union of German Associations of Pharmacists (Other)
Collaborators: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PHARM-CHF
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; medication adherence; pharmacy; interdisciplinary care; randomized controlled trial; mortality; hospitalization
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- regular, pharmacy-based intervention (Experimental): providing medication in weekly dosing aids and regular contacts with the local pharmacy
  Interventions: Behavioral: Regular, pharmacy based intervention
- usual care (No Intervention): usual care

INTERVENTIONS:
Behavioral: Regular, pharmacy based intervention — Regular, pharmacy-based intervention conducted in cooperation with the treating physician:
  * Medication review at baseline: recording of all medicines currently taken (prescribed medication and self-medication), check for drug-related problems, consolidation of a medication plan.
  * Regularly (weekly): dose-dispensing of the medication (weekly dosing aid), discussion and counseling regarding medication, adherence, potential side effects, and signs and symptoms of cardiac decompensation; blood pressure and pulse measurement. If required: contact with patients' physician.
  Arms: regular, pharmacy-based intervention

SUMMARY:
The aim of the study is to investigate whether a continuous interdisciplinary intervention improves medication adherence (primary efficacy endpoint) and leads to a reduction of hospitalizations and mortality (primary safety endpoint) in elderly patients with chronic heart failure. The intervention, consisting of regular contacts with the local pharmacy and weekly dosing aids, aims to improve medication adherence and management.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 years and older
* Chronic heart failure (CHF)
* Stable CHF medication including a diuretic
* Hospitalization for decompensated heart failure within past 12 months OR a value of ≥ 350 pg/mL for BNP or ≥ 1,400 pg/mL for NT-proBNP
* Written informed consent

Exclusion Criteria:

* Use of a weekly dosing aid
* Unwillingness or inability to visit a participating pharmacy once a week
* Planned cardiac surgery
* Life-expectancy < 6 months
* Unwillingness or inability to comply with the study protocol (including drug abuse or alcohol dependency)
* Participation in other studies (currently or in the last 4 weeks)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schulz, Prof. PhD, Study Chair — Federal Union of German Associations of Pharmacists; Ulrich Laufs, Prof. MD, Study Chair — Universitätsklinikum Leipzig
Locations (1):
- Saarland University, Homburg/Saar, Germany

REFERENCES:
- [Derived] Laufs U, Griese-Mammen N, Krueger K, Wachter A, Anker SD, Koehler F, Rettig-Ewen V, Botermann L, Strauch D, Trenk D, Bohm M, Schulz M. PHARMacy-based interdisciplinary program for patients with Chronic Heart Failure (PHARM-CHF): rationale and design of a randomized controlled trial, and results of the pilot study. Eur J Heart Fail. 2018 Sep;20(9):1350-1359. doi: 10.1002/ejhf.1213. Epub 2018 May 30. PMID 29846031
- See also: PHARM-CHF study home page — http://www.pharm-chf.de

RESULTS

PARTICIPANT FLOW:
Groups:
- Regular, Pharmacy-based Intervention: providing medication in weekly dosing aids and regular contacts with the local pharmacy
  Regular, pharmacy based intervention: Regular, pharmacy-based intervention conducted in cooperation with the treating physician:
  * Medication review at baseline: recording of all medicines currently taken (prescribed medication and self-medication), check for drug-related problems, consolidation of a medication plan.
  * Regularly (weekly): dose-dispensing of the medication (weekly dosing aid), discussion and counseling regarding medication, adherence, potential side effects, and signs and symptoms of cardiac decompensation; blood pressure and pulse measurement. If required: contact with patients' physician.
- Usual Care: usual care; no medication review, no dose dispensing; study pharmacists unaware of patients in this group.
Period: Overall Study
Arm/Group | Regular, Pharmacy-based Intervention | Usual Care
Started | 130 | 128
Completed | 110 | 127
Not Completed | 20 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Intervention: pts. did not present to participating pharmacy | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular, Pharmacy-based Intervention | Usual Care | Total
Number analyzed (Participants) | 110 | 127 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (6.8) | 74.1 (7.2) | 74.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 49 | 91
  Male | 68 | 78 | 146
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Percentage of days covered (PDC) by prescribed medication and according to claims data
Time Frame: 12 months
Population: Patients for whom we were able to calculate a PDC.
Measure: Mean (Standard Deviation); unit: percentage of days covered
Arm/Group | Regular, Pharmacy-based Intervention | Usual Care
Number analyzed (Participants) | 90 | 112
percentage of days covered | 91.2 (11.9) | 85.5 (16.6)

2. Primary Outcome: Days Lost Due to Unplanned Cardiovascular Hospitalizations or Death of Any Cause
Description: Days lost due to unplanned cardiovascular hospitalizations or death of any cause
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: days lost
Arm/Group | Regular, Pharmacy-based Intervention | Usual Care
Number analyzed (Participants) | 110 | 127
days lost | 24.8 [10.6 to 38.9] | 16.5 [6.1 to 26.8]

ADVERSE EVENTS:
Time Frame: 365 days and until end of the study
Arm/Group | Regular, Pharmacy-based Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 8/110 | 8/127
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/127
Other Adverse Events (participants affected / at risk) | 0/110 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT01692119/SAP_000.pdf
  • Study Protocol (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT01692119/Prot_001.pdf